CLINICAL TRIAL: NCT03614741
Title: Efficacy, Safety and Pharmacokinetics of Tinzaparin During Slow Low Efficient Daily Dialysis in Intensive Care Patients
Acronym: Tinza-SLEDD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R18098M
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Acute Kidney Injury; Renal Replacement Therapy; Anticoagulants
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Bolus of 4500 IU tinzaparin
  Interventions: Drug: Tinzaparin bolus
- Study group (Active Comparator): Bolus of 4500 IU tinzaparin and continuous infusion of 4500 IU tinzaparin
  Interventions: Drug: Tinzaparin continuous infusion; Drug: Tinzaparin bolus

INTERVENTIONS:
Drug: Tinzaparin continuous infusion — 4500 IU continuous infusion of Tinzaparin
  Arms: Study group
Drug: Tinzaparin bolus — 4500 IU bolus of Tinzaparin

SUMMARY:
This study evaluates the pharmacokinetics of tinzaparin during renal replacement therapy (RRT).

60 patients with clinical indication for pharmacological thromboprophylaxis and slow low efficient daily dialysis (SLEDD) will be studied in Tampere University Hospital. All subjects will receive a 4500 IU bolus of tinzaparin. The subjects in study group (n=30) will also receive a 4500 IU continuous infusion of tinzaparin.

DETAILED DESCRIPTION:
After written informed consent, 60 subjects with clinical indication for pharmacological thromboprophylaxis and SLEDD will be studied in the Tampere University Hospital intensive care unit. After inclusion the subjects will be randomly assigned into study group (30 patients) and control (30 patients).

All subjects receive a bolus of tinzaparin 4500 IU into the inlet line of dialyzer at 5 minutes after the start of blood pump. Afterwards the subjects in the study group will continue to receive continuous tinzaparin infusion (concentration 100 IU/ml) 500 IU/h over seven hours. No other heparin product (including arteria flush lines) nor dilution fluids at the dialyzer are allowed during the study period of 24 hours. Each SLEDD treatment will be performed with Cordiax 5008S (Fresenius) for 8 hours. After the study period of 24 hours thromboprophylaxis will be prescribed according to the normal practice in the ICU.

The primary outcome measure is plasma anti-FXa concentration at 4 hours from the onset of SLEDD. Plasma Anti-FXa will be drawn at timepoints 0 hours, 4 hours, 8 hours and 24 hours from the onset of the dialysis.

The clotting formation in RRT system will be evaluated by clotting scoring. In the case of serious clotting RRT treatment is stopped and the new RRT is started. The study will end to the new RRT.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients requiring intensive care
* Indication for pharmacological thromboprophylaxis
* Written informed consent obtained from the patient or his/her legal representative
* Indication for SLEDD, any of following:
* serum creatinine concentration of more than 354 micromol/l or greater than 3 times the baseline creatinine level OR
* anuria (urine output of 100 ml/day) for more than 12 hours OR
* oliguria: below 0.3 ml/kg/h for more than 24 hours OR 500 ml/day
* the presence of clinically significant organ edema (e.g., pulmonary edema, elevated intra-abdominal pressure, significant peripheral swelling) together with oliguria or anuria
* Dialysis dependence after continuous renal replacement treatment

Exclusion Criteria:

* Other indications for anticoagulant therapy than thromboprophylaxis (including sodium citrate for CRRT)
* Any long-term anticoagulant or antithrombotic medication, except for low-dose aspirin (<150 mg daily)
* Treatment with tinzaparin or any other LMWH or heparin within 24 hours of study inclusion
* Known heparin induced thrombocytopenia (HIT), or hypersensitivity to tinzaparin or any other heparin
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma anti-FXa concentration | 4 hours from the onset of SLEDD
  Plasma anti-factor Xa blood sample

SECONDARY OUTCOMES:
Plasma anti-FXa concentration | 8 hours from the onset of SLEDD
  Plasma anti-factor Xa blood sample
Plasma anti-FXa concentration | 24 hours from the onset of SLEDD
  Plasma anti-factor Xa blood sample
Clotting Score | 8 hours from the onset of SLEDD
  Clotting in renal replacement sircuit will be evaluated hourly according to predescribed score

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kuitunen, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No